CLINICAL TRIAL: NCT06352255
Title: Analysis of Pain and Anxiety With Carpule vs Syringe in Digital Anesthesia of the Hallux
Brief Title: Pain and Anxiety During Local Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, ANA MARIA RAYO PEREZ, Principal Investigator, University of Seville
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: AR1937
Record Dates: First submitted 2023-10-26; First posted 2024-04-08 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Anesthesia, Local; Pain; Anxiety
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital block with carpule. (Experimental): The study group will be made up of subjects who will undergo anesthetic block with carpule.
  Interventions: Procedure: Digital block
- Digital block with syringe. (Active Comparator): The control group will be made up of the subjects who will undergo anesthetic block with syringe.
  Interventions: Procedure: Digital block

INTERVENTIONS:
Procedure: Digital block — Frost's H technique

SUMMARY:
INTRODUCTION: Currently, there is no scientific evidence about pain in the anesthetic blockage of the first finger according to the application method. However, clinical evidence has valued the use of carpule, due to the low pain it generates in the patient to the application of anesthetic. Most studies on anesthesia and pain, especially with the use of carpule and distracting methods, belong to the field of dentistry.

OBJECTIVES: It is intended to determine the pain after an anesthetic block in H of Frost in the first finger with different application methods, such as syringe and carpule. As secondary objectives, it is intended to establish the difference in pain according to the sex and age of the patients.

METHODOLOGY: Experimental, transverse and random clinical trial type analytical study, in which a sample of 200 individuals will be selected, 100 per group, which would require digital anesthesia of the first finger and that would fulfill the inclusion criteria.

Result: after the completion of the study CONCLUSIONS: After the completion of the study

ELIGIBILITY:
Inclusion Criteria:

* Subjects over 18 years of age
* Both sexes
* Participants must present nail pathology that requires surgical intervention.

Exclusion Criteria:

* Systemic degenerative
* Neuromuscular diseases
* Pregnant or likely to be pregnant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-07-20 (Actual)

PRIMARY OUTCOMES:
Grade of Pain postinyection | Immediately after the intervention
  Analyze the pain using the VAS scale (Visual Analog Scale) caused during the anesthetic process. The lowest score on this scale is 0 (no pain) and the highest is 10 (maximum bearable pain).

SECONDARY OUTCOMES:
Anxiety before the intervention | Immediately before the intervention, since it is a scale that scores from 1 to 3 the degree of anxiety of the patient prior to the surgical intervention.
  Compare the degree of anxiety of patients undergoing the anesthetic procedure using syringe vs carpule.

CONTACTS AND LOCATIONS:
Overall Officials: ANA M RAYO PEREZ, Doctor, Principal Investigator — University of Seville
Locations (1):
- Clinica Rayo, Seville, Spain

IPD SHARING:
Plan to Share IPD: No